CLINICAL TRIAL: NCT03549416
Title: BioDay Registry: Prospective, Observational Data Collection Regarding the Use of New Systemic Treatment Options in Patients with Atopic Diseases in Daily Practice
Brief Title: BioDay Registry: Data Collection Regarding the Use of New Systemic Treatment Options in Patients with Atopic Dermatitis
Acronym: BioDay
Status: Recruiting | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: Academisch Ziekenhuis Groningen (Other); Sanofi (Industry); AbbVie (Industry); Eli Lilly and Company (Industry); LEO Pharma (Industry)
Responsible Party: Principal Investigator, Dr M.S. de Bruin-Weller, M.S. de Bruin-Weller, dermatologist, MD, PhD, UMC Utrecht
Other Study IDs: 18/239
Record Dates: First submitted 2018-05-25; First posted 2018-06-08 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; Dupilumab; Dupixent; BioDay; Daily practice; Real world; Atopic Diseases Registry; Registry; Multi center; Biologics; Janus kinase inhibitors; Baricitinib; Upadacitinib; Abrocitinib; Tralokinumab
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The BioDay Registry aims to address the need for daily practice data regarding the effectiveness and safety of new systemic treatment options (like biologics and Janus kinase inhibitors) in patients with atopic dermatitis and effect on other atopic comorbidities in a multicenter setting. The registry already consists of several additional modules concerning atopic comorbidities, like food allergy and asthma, and a module for conjunctivitis during biologic treatment.

ELIGIBILITY:
Inclusion Criteria:

* All adult and paediatric patients treated with new systemic treatments for AD will be asked for participation in the BioDay Registry

Exclusion Criteria:

* Patients are not eligible for enrolment in case of presumed inability to answer questionnaires or not willing to answer questionnaires and will be excluded.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All adult and paediatric patients treated with new systemic treatments for AD will be asked for participation in the BioDay Registry
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of effectiveness | Change from baseline to previous specified timepoints (16 weeks, 1 year, 2 year etc.)
  To assess the effectiveness of new treatments in adult and pediatric patients with AD using physician measured clinical eczema scores as well as patient-reported outcome measures.
Drug survival | Drug survival analysis, which is the length of time a patient continues to take a particular drug, will be performed every year, with cumulative results over the years.
  To study drug survival and identify factors that affect drug survival.
Side effects | Change from baseline to previous specified timepoints (16 weeks, 1 year, 2 year etc.)
  To register objective and subjective side effects and to identify potential risk factors.

SECONDARY OUTCOMES:
Characterization of population | Yearly from baseline up to 5 years
  To characterize patient populations treated with new AD treatments in daily practice.
Characterization of side effects | Yearly from baseline up to 5 years
  To collect data from daily practice regarding side effects (incidence, severity, risk factors, treatment options, etc.).
Laboratory monitoring | Yearly from baseline up to 5 years
  To study the usefulness of laboratory monitoring during treatment in daily practice, with emphasis on subpopulations (e.g. elderly patients, patients with pre-existing liver and/or renal disease).
Long-term safety | Yearly from baseline up to 5 years
  To study the long-term safety risks including malignancies, pregnancy/paternity-related conditions, infections, and autoimmune diseases.
Comorbidities | Yearly from baseline up to 5 years
  To prospectively collect data from daily practice regarding the effect of new treatment options for AD on comorbidities (for example atopic diseases like asthma, food allergy and rhinoconjunctivitis can improve from these new drugs as many target the Th2 axis).
Dose tapering | Yearly from baseline up to 5 years
  To assess whether dose reduction of biologics can be achieved in patients with low AD activity.

CONTACTS AND LOCATIONS:
Overall Officials: Marjolein de Bruin-Weller, Md, PhD, Principal Investigator — UMC Utrecht
Locations (14):
- Netherlands (14):
  - Radboud University Medical Center, Nijmegen, Gelderland
  - Isala Dermatologisch Centrum, Zwolle, Overijssel
  - Medisch Centrum Leeuwarden, Leeuwarden, Provincie Friesland
  - University Medical Center Groningen, Groningen, Provincie Groningen
  - IJsselland Ziekenhuis, Capelle aan den IJssel, South Holland
  - University Medical Center Utrecht, Utrecht, Utrecht
  - Meander Medisch Centrum, Amersfoort
  - Reinier de Graaf ziekenhuis, Delft
  - Catharina ziekenhuis, Eindhoven
  - Spaarne Gasthuis, Haarlem
  - Maastricht Univeristy Medical Center, Maastricht
  - Haga ziekenhuis, The Hague
  - Diakonessenhuis, Utrecht
  - St Antonius ziekenhuis, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clabbers J, Boesjes C, Spekhorst L, van Gisbergen MW, Maas E, Marshall J, Janssen R, Janssen M, Zuithoff N, Steijlen P, de Graaf M, van Geel M, de Bruin-Weller M, Gostynski A. Influence of pathogenic filaggrin variants on dupilumab treatment in atopic dermatitis. J Allergy Clin Immunol. 2024 Apr;153(4):1155-1161.e4. doi: 10.1016/j.jaci.2023.12.027. Epub 2024 Jan 23. PMID 38272373